CLINICAL TRIAL: NCT00824486
Title: A Randomized Trial of a Home Safety Intervention Using a Safe Home Model
Brief Title: Home Safety Intervention Using a Safe Home Model
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Elizabeth C. Powell, MD, MPH, Children's Memorial Hospital
Allocation: Randomized | Model: Single Group
Other Study IDs: 2003-12084
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Last update posted 2009-01-16 (Estimated); Status verified 2009-01

CONDITIONS: Healthy
Keywords: child; injury prevention
MeSH Terms: interventions — tyrosyl-1,2,3,4-tetrahydro-3-isoquinolinecarbonyl-phenylalanyl-phenylalanine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TIPP (Active Comparator): Injury prevention education using TIPP materials
  Interventions: Behavioral: Injury prevention education (TIPP)
- Safe Home Model (Experimental): Injury prevention education using safe home model
  Interventions: Behavioral: Injury prevention education (safe home)

INTERVENTIONS:
Behavioral: Injury prevention education (TIPP) — using TIPP materials
  Arms: TIPP
Behavioral: Injury prevention education (safe home) — using safe home model
  Arms: Safe Home Model

SUMMARY:
This project seeks to determine the efficacy of safety education using a safe home model. The 4 X 8 ft. model is designed to look like a house; each of 4 "rooms" has a focused safety message. Families will be enrolled in the clinic and randomized to one of two groups, the safe home model group and the printed safety education materials (TIPP materials) group. The investigators will compare the retention of safety information among caregivers instructed using these two methods. The hypothesis is that families in the safe home model group will have improved retention of safety information.

ELIGIBILITY:
Inclusion Criteria:

* Caregivers of children younger than 6 years old

Exclusion Criteria:

* Language other than English or Spanish

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-06; Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Memorial Hospital, Chicago, Illinois, United States